CLINICAL TRIAL: NCT05795504
Title: Resistive Exercise Versus High Intensity Interval Training on Calcium and Vitamin D in Premenopausal Women: A Randomized Controlled Trial
Brief Title: Resistive Exercise Versus HIIT on Calcium and Vitamin D
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Mohamed Ali Shehata, lecturer of physical therapy for women's health, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P.T.REC/012/004342
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Vitamin D Deficiency; Calcium; Premenopause
MeSH Terms: conditions — Vitamin D Deficiency | interventions — High-Intensity Interval Training; Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- resistive exercises (Experimental): Premenopausal women in group A will perform resistive exercise for upper and lower limbs, three times per week in addition to calcium and vitamin d supplementations.
  Interventions: Other: resistive exercise; Dietary Supplement: calcium and vitamin D
- high intensity interval training (Experimental): Premenopausal women in group B will receive high intensity interval training for three times per week in addition to calcium and vitamin D supplementations
  Interventions: Other: high intensity interval training; Dietary Supplement: calcium and vitamin D
- conventional therapy (Active Comparator): Premenopausal women in group C will receive calcium and vitamin D supplementations only.
  Interventions: Dietary Supplement: calcium and vitamin D

INTERVENTIONS:
Other: resistive exercise — They will perform combined upper and lower resistive exercises, 30 min, 3 sessions / week for 12 weeks in addition to calcium and vitamin D supplements.
  Arms: resistive exercises
Other: high intensity interval training — They will perform HIIT for three sessions/ week for 12 weeks, 30 minutes/ session in addition to calcium and vitamin D supplements.,
  Arms: high intensity interval training
Dietary Supplement: calcium and vitamin D — they will receive calcium and vitamin D supplements only.

SUMMARY:
A comparison between resistive exercise and high intensity interval trainig on calcium and vitamin d in premenopausal women.

DETAILED DESCRIPTION:
A total of 57% of women were vitamin D deficient with higher vitamin D deficiency found among premenopausal women (64.7%). Concentrations of 25(OH) D, defined as severely deficient (< 12 ng/ml), deficient (12-19 ng/ml), insufficient (20-30 ng/ml) and sufficient (> 30 ng/ml). Both severe vitamin D deficiency and calcium deficiency was significantly more frequent in premenopausal women compared to postmenopausal women. So, it is important to find effective therapeutic approaches to treat vitamin D deficiency among these women

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women having reduced calcium level (less than 500mg) intake as recorded by 24 hours' dietary recall method and vitamin D deficiency (12-19 ng/ml).
* Their ages will range from 40 to 45 years.
* Their BMI will range from 25-30 kg/m2.
* Don't receive hormonal replacement therapy.

Exclusion Criteria:

* Smoking.
* History of chronic disease (uncontrolled hypertension, diabetes mellitus)
* Osteoporosis.
* severe musculoskeletal disorders
* cardiovascular disease, thyroid dysfunction

Ages: 40 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Vitamin D serum level | three months
  a blood sample of each participant will be taken to measure serum vitamin D level before and after the study
serum calcium level | three months
  a blood sample will be taken from each participant to measure calcium level of each participant before and after the study.

CONTACTS AND LOCATIONS:
Overall Officials: Mai shehata, Principal Investigator — faculty of physical therapy
Locations (1):
- Faculty of physical therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No